CLINICAL TRIAL: NCT03250819
Title: Genetic Association Study on Corticosteroid-induced Elevation of the Intraocular Pressure
Brief Title: Gene Polymorphisms of Corticosteroid-induced Ocular Hypertension
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL58992.068.17
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Corticosteroid Induced Ocular Hypertension/Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Corticosteroid responders: Patients who develop an increase in eye pressure after the use of corticosteroids
  Interventions: Other: SNP analysis
- Non-corticosteroid responders: Patients who use/used corticosteroids but didn't develop an increase in eye pressure
  Interventions: Other: SNP analysis

INTERVENTIONS:
Other: SNP analysis — The collected blood samples will be used to investigate the occurrence of SNPs (single nucleotide polymorphisms) in both study groups

SUMMARY:
Glaucoma is one of the most prevalent eye diseases and the second most common cause of blindness worldwide. The most common form is primary open angle glaucoma (POAG). Glaucoma is a slowly progressing neuropathy of the optic nerve that causes loss of visual field and eventually blindness. Elevated intra-ocular pressure (IOP) is the most important risk factor.

Corticosteroids, which are often used for the treatment of many diseases in ophthalmology and other specialities, may cause an elevation of the IOP. It is estimated that corticosteroids induce ocular hypertension in approximately 18%-36% of the general population and in patients with POAG this percentage can be as high as 92%. When the treatment is sustained, this can cause a glaucomatous neuropathy of the optic nerve (corticosteroid-induced glaucoma).

The precise pathogenic mechanism isn't clear yet. Genetic factors are likely to affect the susceptibility to corticosteroid response. Therefore, an overview of the genetic mechanisms of corticosteroid-induced glaucoma can give more insight in the pathogenesis. In this study the researchers investigate the occurrence of SNPs (single nucleotide polymorphisms) in 150 cases with a steroid-response in comparison with 300 controls exposed to corticosteroids without a steroid-response.

Up to now, one small GWAS has been conducted comparing 32 patients with and without corticosteroid-induced ocular hypertension after treatment with intravitreal triamcinolone. In this study, two SNPs proximal of the transcriptional start site (near the 5') of HCG22 on chromosome 6 were identified. However, this is a rather small sample population and the investigators didn't match for the underlying disease. Further, in another small study, Hogewind et al. performed SNP analysis in multiple genes (SFRS3, FKBP4, FKBP5, and NR3C1) in corticosteroid-induced ocular hypertension.

This study enables the investigators to identify patients at risk for developing corticosteroid-induced glaucoma and to gain a better insight in the pathogenesis. This may also lead to the discovery of biomarkers that indicate an increased risk of developing a steroid-induced glaucoma and new prevention and treatment strategies, which are necessary as the treatment of corticosteroid induced-glaucoma now only focuses at lowering the IOP and can still be challenging.

ELIGIBILITY:
Inclusion Criteria:

* Use of corticosteroids:
* Patients treated with Ozurdex (an intravitreal dexamethasone implant
* Patients treated with subconjunctival Triamcinolone/ Celestone injections
* Patients treated with corticosteroids after a corneal surgery
* Patients treated with corticosteroids after a refractive surgery
* Patients treated with corticosteroids after a cataract surgery
* Patients treated with corticosteroids for macular edema
* Patients exposed to corticosteroids for other diseases such as uveitis
* When using topical corticosteroids, time of use > 3 months
* Age > 18 year and mentally competent
* Patient from the Maastricht University Medical Centre+ (MUMC+), the Netherlands

Exclusion Criteria:

* Age < 18 year
* Mentally not able to participate or give permission
* Not able to communicate in Dutch
* Patients with a type of uveitis that might cause a decrease of the IOP
* When using topical corticosteroids, time of use < 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who started topical, intravitreal or subconjunctival corticosteroids will be included at the University Eye Clinic Maastricht of the Maastricht University Medical Centre+, the Netherlands. The participants will be divided in two groups: cases who are corticosteroid responder (n=150) and controls exposed to corticosteroids who did not respond with an IOP increase (n=300).
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Differences in SNP's in corticosteroid responders and non-responders | At the time of inclusion
  What are the differences in SNPs in patients with corticosteroid-induced ocular hypertension in comparison with patients exposed to corticosteroids who do not respond with an IOP increase

CONTACTS AND LOCATIONS:
Overall Officials: Johannes SA Schouten, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- University Eye Clinic Maastricht, Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jeong S, Patel N, Edlund CK, Hartiala J, Hazelett DJ, Itakura T, Wu PC, Avery RL, Davis JL, Flynn HW, Lalwani G, Puliafito CA, Wafapoor H, Hijikata M, Keicho N, Gao X, Argueso P, Allayee H, Coetzee GA, Pletcher MT, Conti DV, Schwartz SG, Eaton AM, Fini ME. Identification of a Novel Mucin Gene HCG22 Associated With Steroid-Induced Ocular Hypertension. Invest Ophthalmol Vis Sci. 2015 Apr;56(4):2737-48. doi: 10.1167/iovs.14-14803. PMID 25813999
- [Background] Fini ME, Schwartz SG, Gao X, Jeong S, Patel N, Itakura T, Price MO, Price FW Jr, Varma R, Stamer WD. Steroid-induced ocular hypertension/glaucoma: Focus on pharmacogenomics and implications for precision medicine. Prog Retin Eye Res. 2017 Jan;56:58-83. doi: 10.1016/j.preteyeres.2016.09.003. Epub 2016 Sep 22. PMID 27666015